CLINICAL TRIAL: NCT03949140
Title: Laser Hair Removal for Primary Treatment of Pilonidal Disease Requiring Surgical Intervention
Brief Title: Laser Hair Removal for Treatment of Pilonidal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Syneron Candela (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-1031; Protocol Version 6 (Other: UW Madison); A539790 (Other: UW Madison); SMPH/SURGERY/PEDIATRIC SURGERY (Other: UW Madison)
Record Dates: First submitted 2018-11-16; First posted 2019-05-14 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Pilonidal Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laser hair removal treatment (Experimental): Patients who choose to enroll will plan to undergo a total of up to 8 laser hair removal sessions every 4-6 weeks. If patients develop abscess or infection during this time, they will undergo I&D and/or antibiotics, consistent with standard therapy for infection or abscess. If patients have 2 or more infections in 1 year, pain or drainage for more than 1 month, or miss more than 1 week of school or work due to ineffective treatment of pilonidal disease, these patients will undergo surgical excision and subsequent follow-up at surgeon's discretion. Patients will follow up at 2-4-week intervals for 3 months, then at 6, 9, and 18 months after conclusion of the laser therapy sessions. At all follow-up sessions, patients will be given the DQLI, CDQLI, and Promis 3A Pain survey. Unscheduled visits such as unplanned clinic visits, emergency department encounters, and hospitalizations, will be included in data collected for analysis of primary and secondary outcomes.
  Interventions: Procedure: Laser hair removal

INTERVENTIONS:
Procedure: Laser hair removal — Those who consent to participate in the study will be treated with up to 8 sessions of laser hair removal utilizing a long-pulsed laser to the natal cleft at treatment intervals of 4-6 weeks.
  Other Names: Laser depilation

SUMMARY:
This project is a pilot study to determine if symptomatic pilonidal disease can be primarily managed with laser hair removal vs surgery.

DETAILED DESCRIPTION:
This project will consist of surgical evaluation in pediatric surgery or colorectal surgery clinics, referral to dermatology clinic for informed consent, and if enrolled, participation in up to 8 laser hair removal sessions with regular follow-up for a period of 2 years after completion of therapy.

ELIGIBILITY:
Inclusion Criteria:

Patients with symptomatic pilonidal disease, who meet criteria for surgical intervention:

* Experience two or more episodes of infection or abscess in the past 12 months
* Have pain or drainage for a total of more than 1 month in the past 12 months
* Missed a total of more than 1 week of school or work in the past 12 months
* English-speaking

Exclusion Criteria:

* Patients who have co-morbidities that prevent them from becoming a surgical candidate

  * Previous history of laser hair removal in the gluteal cleft (prior to initial enrollment)
  * Previous excision of pilonidal sinus (prior to initial enrollment)
  * Non-English speaking

Ages: 13 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Incidence of disease-free remission | up to 2 years
  Disease free rate among those subjects who only required laser therapy. Disease-free remission will be assessed at 12 and 24 months.
Disease recurrence rate among subjects who subsequently require surgical intervention. | up to 2 years
  Rate of recurrence of pilonidal disease among subjects who participated in the study but also required surgical intervention.

SECONDARY OUTCOMES:
Characterization of the degree of intervention required to obtain positive results. | up to 2 years
  Incision and drainage vs. need for larger excision, requirement for oral antibiotics, and the number of emergency room visits, or hospital admissions related to pilonidal disease.
Number of missed school or work days | Up to 18 months
  This study will investigate qualitative outcomes including the number of missed school or work days at each follow up, 6, 9, and 18 months.
Assessment of Pain via Promis 3A Pain Short Form | up to 18 months
  This study will investigate qualitative outcomes including pain. Pain will be assessed via the Promis 3A Pain Short Form at 6, 9, and 18 months. This is a one question survey that has participants rate the intensity of their pain over the last 7 days, on average. The scale is from 0-10 where 0 is no pain and 10 is the worst pain imaginable.
Number of Days Participants Experience Drainage | up to 18 months
  This study will investigate qualitative outcomes including assessment of drainage. This will be reported as the number of days participants experienced drainage since last follow up, assessed at 6, 9, and 18 month follow up.
Cost-benefit analysis of laser hair-treated patients versus matched historical control. | up to 2 years
  Evaluate total cost to the health care system relative to period of disease-free remission.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] von Laffert M, Stadie V, Ulrich J, Marsch WC, Wohlrab J. Morphology of pilonidal sinus disease: some evidence of its being a unilocalized type of hidradenitis suppurativa. Dermatology. 2011;223(4):349-55. doi: 10.1159/000335373. Epub 2012 Jan 21. PMID 22269798
- [Background] Sondenaa K, Pollard ML. Histology of chronic pilonidal sinus. APMIS. 1995 Apr;103(4):267-72. doi: 10.1111/j.1699-0463.1995.tb01105.x. PMID 7542011
- [Background] Sondenaa K, Andersen E, Nesvik I, Soreide JA. Patient characteristics and symptoms in chronic pilonidal sinus disease. Int J Colorectal Dis. 1995;10(1):39-42. doi: 10.1007/BF00337585. PMID 7745322
- [Background] Al-Khamis A, McCallum I, King PM, Bruce J. Healing by primary versus secondary intention after surgical treatment for pilonidal sinus. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD006213. doi: 10.1002/14651858.CD006213.pub3. PMID 20091589
- [Background] Steele SR, Perry WB, Mills S, Buie WD; Standards Practice Task Force of the American Society of Colon and Rectal Surgeons. Practice parameters for the management of pilonidal disease. Dis Colon Rectum. 2013 Sep;56(9):1021-7. doi: 10.1097/DCR.0b013e31829d2616. No abstract available. PMID 23929010
- [Background] Stauffer VK, Luedi MM, Kauf P, Schmid M, Diekmann M, Wieferich K, Schnuriger B, Doll D. Common surgical procedures in pilonidal sinus disease: A meta-analysis, merged data analysis, and comprehensive study on recurrence. Sci Rep. 2018 Feb 15;8(1):3058. doi: 10.1038/s41598-018-20143-4. PMID 29449548
- [Background] Doll D, Krueger CM, Schrank S, Dettmann H, Petersen S, Duesel W. Timeline of recurrence after primary and secondary pilonidal sinus surgery. Dis Colon Rectum. 2007 Nov;50(11):1928-34. doi: 10.1007/s10350-007-9031-4. PMID 17874268
- [Background] Khan MA, Javed AA, Govindan KS, Rafiq S, Thomas K, Baker L, Kenealy J. Control of hair growth using long-pulsed alexandrite laser is an efficient and cost effective therapy for patients suffering from recurrent pilonidal disease. Lasers Med Sci. 2016 Jul;31(5):857-62. doi: 10.1007/s10103-016-1920-0. Epub 2016 Mar 22. PMID 27003897
- [Background] Dragoni F, Moretti S, Cannarozzo G, Campolmi P. Treatment of recurrent pilonidal cysts with nd-YAG laser: report of our experience. J Dermatolog Treat. 2018 Feb;29(1):65-67. doi: 10.1080/09546634.2017.1329513. Epub 2017 May 30. PMID 28521574
- [Background] Oram Y, Kahraman F, Karincaoglu Y, Koyuncu E. Evaluation of 60 patients with pilonidal sinus treated with laser epilation after surgery. Dermatol Surg. 2010;36(1):88-91. doi: 10.1111/j.1524-4725.2009.01387.x. Epub 2009 Dec 4. PMID 20002644
- [Background] Pronk AA, Eppink L, Smakman N, Furnee EJB. The effect of hair removal after surgery for sacrococcygeal pilonidal sinus disease: a systematic review of the literature. Tech Coloproctol. 2018 Jan;22(1):7-14. doi: 10.1007/s10151-017-1722-9. Epub 2017 Nov 28. PMID 29185064
- [Background] Toosi P, Sadighha A, Sharifian A, Razavi GM. A comparison study of the efficacy and side effects of different light sources in hair removal. Lasers Med Sci. 2006 Apr;21(1):1-4. doi: 10.1007/s10103-006-0373-2. Epub 2006 Apr 1. PMID 16583183
- [Background] Nanni CA, Alster TS. Laser-assisted hair removal: side effects of Q-switched Nd:YAG, long-pulsed ruby, and alexandrite lasers. J Am Acad Dermatol. 1999 Aug;41(2 Pt 1):165-71. doi: 10.1016/s0190-9622(99)70043-5. PMID 10426883
- [Background] Mutus HM, Aksu B, Uzun E, Gulcin N, Gercel G, Ozatman E, Durakbasa CU, Okur H. Long-term analysis of surgical treatment outcomes in chronic pilonidal sinus disease. J Pediatr Surg. 2018 Feb;53(2):293-294. doi: 10.1016/j.jpedsurg.2017.11.031. Epub 2017 Nov 14. PMID 29217319
- [Background] Pascoe VL, Kimball AB. Seasonal variation of acne and psoriasis: A 3-year study using the Physician Global Assessment severity scale. J Am Acad Dermatol. 2015 Sep;73(3):523-5. doi: 10.1016/j.jaad.2015.06.001. No abstract available. PMID 26282801
- [Background] Kimball AB, Jemec GB, Yang M, Kageleiry A, Signorovitch JE, Okun MM, Gu Y, Wang K, Mulani P, Sundaram M. Assessing the validity, responsiveness and meaningfulness of the Hidradenitis Suppurativa Clinical Response (HiSCR) as the clinical endpoint for hidradenitis suppurativa treatment. Br J Dermatol. 2014 Dec;171(6):1434-42. doi: 10.1111/bjd.13270. Epub 2014 Nov 11. PMID 25040429